CLINICAL TRIAL: NCT05256108
Title: A Single-dose, Randomized, Double-blind, Placebo- and Active-controlled Crossover Trial to Evaluate the Abuse Potential of Two Doses of Cebranopadol in Adult Nondependent Recreational Opioid Users
Brief Title: Assessment of Abuse Potential of Cebranopadol in Humans
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tris Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PARK-101-HAP
Record Dates: First submitted 2022-02-16; First posted 2022-02-25 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-02

CONDITIONS: Human Abuse Potential
Keywords: pain; abuse; opioid
MeSH Terms: conditions — Pain | interventions — Oxycodone; Tramadol; 6'-fluoro-4',9'-dihydro-N,N-dimethyl-4-phenylspiro(cyclohexane-1,1'(3'H)-pyrano(3,4-b)indol)-4-amine

STUDY DESIGN:
Intervention Model Description: Randomized, single site, double-blind, placebo- and active-controlled, crossover, single oral dose, Phase 1 trial, in non dependent recreational opioid users
Who Masked: Participant, Investigator
Masking Description: To ensure blinding to the treatment, subjects will receive 6 identically looking capsules that will contain one of the 5 assigned treatments. Subjects will be randomized 1:1:1:1:1 and will receive one of 2 cebranopadol doses: oxycodone IR: tramadol IR: placebo in each of the 5 treatment periods.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cebranopadol 600 µg (Experimental): Single oral dose of 6 capsules containing 3 cebranopadol 200 µg tablets and placebo
  Interventions: Drug: Cebranopadol 600 µg
- Cebranopadol 1000 µg (Experimental): Single oral dose of 6 capsules containing 5 cebranopadol 200 µg tablets and placebo
  Interventions: Drug: Cebranopadol 1000 µg
- Oxycodone 40 mg (Active Comparator): Single oral dose of 6 capsules containing 2 oxycodone 20 mg and placebo
  Interventions: Drug: Oxycodone 40 mg
- Tramadol 600 mg (Active Comparator): Single oral dose of 6 capsules containing 6 tramadol 100 mg tablets
  Interventions: Drug: Tramadol 600 mg
- Placebo (Placebo Comparator): Single oral dose of 6 capsules containing placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxycodone 40 mg — Participants will be administered a single dose of 6 capsules containing oxycodone and placebo in a randomized crossover manner
  Other Names: Qualification Phase/ Treatment Phase
  Arms: Oxycodone 40 mg
Drug: Tramadol 600 mg — Participants will be administered a single dose of 6 capsules containing tramadol in a randomized crossover manner
  Other Names: Qualification Phase/ Treatment Phase
  Arms: Tramadol 600 mg
Drug: Placebo — Participants will be administered a single dose of 6 capsules containing placebo in a randomized crossover manner
  Other Names: Qualification Phase/ Treatment Phase
  Arms: Placebo
Drug: Cebranopadol 600 µg — Participants will be administered a single dose of 6 capsules containing cebranopadol and placebo in a randomized crossover manner
  Other Names: Treatment Phase
  Arms: Cebranopadol 600 µg
Drug: Cebranopadol 1000 µg — Participants will be administered a single dose of 6 capsules containing cebranopadol and placebo in a randomized crossover manner
  Other Names: Treatment Phase
  Arms: Cebranopadol 1000 µg

SUMMARY:
This study will be conducted to evaluate the abuse potential of single doses of cebranopadol as compared with oxycodone, tramadol and matching placebo in recreational drug users.

DETAILED DESCRIPTION:
Randomized, single site, double-blind, placebo- and active-controlled, crossover, single oral dose, Phase 1 trial, in non dependent recreational opioid users

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent
* Adult men or women aged 18 to 55 years, inclusive
* History of recreational opioid use defined as non therapeutic use at least 10 times in the subject's lifetime and at least once in the 12 weeks prior to the Enrollment Visit
* Body mass index between 19 kg/m2 and 32 kg/m2 inclusive, with a body weight of not less than 50 kg at Enrollment
* Subjects must be in good health as determined by medical history, physical examination, 12 lead electrocardiogram (ECG), and vital signs (pulse rate, systolic blood pressure and diastolic blood pressure, respiratory rate, and oxygen saturation using pulse oximetry) at Enrollment

Exclusion Criteria:

* Exclusion Criteria for Enrollment:
* Self-reported history of drug or alcohol dependence (lifetime) other than caffeine or nicotine as defined by DSM IV-TR criteria
* Current treatment or treatment within their lifetime for substance disorders, other than treatment for smoking cessation
* Positive or missing alcohol breath test at Enrollment; the alcohol breath test can be repeated and/or the subject rescheduled at the discretion of the investigator or designee
* Pregnant or breastfeeding or missing pregnancy test
* Unwillingness or inability to abstain from recreational drug use for the duration of the trial
* Current consumption of greater than 20 cigarettes per day or inability to abstain from smoking (or use of any nicotine-containing substance) for at least 8 hours
* Participation in another clinical trial within 30 days prior to Enrollment that resulted in the administration of at least 1 dose of IMP
* Diseases or conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs. Subjects with a history of cholecystectomy are not excluded
* Prolongation of QTcF (after repeated assessment) at Enrollment, i.e., >450 ms for men or >470 ms for women, or presence of additional risk factors for torsade de pointes (e.g., heart failure, hypokalemia), or use of concomitant medications that prolong the QT interval
* History of orthostatic hypotension or other cardiovascular diseases
* Any clinically significant disease that in the investigator's opinion may affect efficacy or safety assessments or may compromise the subject's safety during trial participation, e.g., significant pulmonary, gastrointestinal, cardiac, endocrine, metabolic, neurological, or psychiatric disorders
* Definite or suspected history of drug allergy or hypersensitivity to opioids or opioid antagonists
* Use of prescription medications within the longer of 14 days or 5 half-lives or use of over-the-counter medications within the longer of 7 days or 5 half-lives prior to dosing, exceptions may be made on a case-by-case basis (e.g., for medications with a short half-life or for topical medications) if approved by the medical monitor in agreement with the investigator
* Any contraindication for naloxone, oxycodone IR, or tramadol IR administration
* Not able to abstain from consumption of beverages or food containing caffeine (tea, coffee, cola, chocolate, etc.) or alcohol from 2 days prior to each Day 1 until discharge from the research unit; beverages or food containing quinine (e.g., bitter lemon, tonic water) from 1 week before Day 1 of the Qualification Phase until the final examination; grapefruit juice (sweet or sour) or Seville oranges from 1 week before Day 1 of the Qualification Phase until the final examination.
* Blood loss of 500 mL or more within 4 weeks before dosing in the treatment phase in this trial, including blood donation. Planned blood donations during the trial and up to 12 weeks after the Final Examination
* History of seizure disorder including unprovoked seizure and/or epilepsy or any condition associated with a significant risk for seizure disorder or epilepsy at the Enrollment Visit at the discretion of the investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2022-07-12 (Actual)

PRIMARY OUTCOMES:
Drug Liking Visual analog scale (VAS) Emax | Treatment Phase: Intervals from predose to 48 hours post-dose
  The scale is a 0-100-point scale: 0 = "Strong disliking"; 50 = "Neither like nor dislike"; 100 = "Strong liking"

SECONDARY OUTCOMES:
VAS rating for Overall Liking | Treatment Phase: Intervals from predose to 48 hours post-dose
  The scale is a 0-100-point scale: 0 = "Strong Disliking", 50 = "Neither Like nor Dislike", 100 = "Strong Liking"
VAS rating for Take Drug Again | Treatment Phase: Intervals from predose to 48 hours post-dose
  The scale is a 0-100-point scale: 0 = "Definitely would not"; 50 = "Do not care"; 100 = "Definitely would"
Pupillometry | Treatment Phase: Intervals from predose to 48 hours post-dose
  Data from a series of frames will be used in the calculation, and the final display will show the weighted average and standard deviation of the pupil size. Measurements will be collected under mesopic lighting conditions
Multi-Tasking Test | Treatment Phase: Intervals from predose to 48 hours post-dose
  Formerly known as the Attention Switching Task (AST), is a test of executive function which provides a measure of the ability to use multiple sources of potentially conflicting information to guide behavior.

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio Clinical Trials, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No